CLINICAL TRIAL: NCT07080151
Title: Zhongshan Hospital Cardiovascular Imaging Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Head of Department of Cardiology, Shanghai Zhongshan Hospital
Other Study IDs: ZSCD2025
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Atherosclerosis; Cardiovascular Diseases
Keywords: Computed Tomography Angiography; Coronary Angiography; Intravascular Ultrasound; Optical Coherence Tomography; Cardiac Magnetic Resonance Imaging
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study cohort: Patients who underwent CAG or CTA during Aug 1st, 2025 and Dec 31st, 2035 at Zhongshan Hospital will be included in this registry. In addition, patients with CTA or at least one of OCT/IVUS/CMR between Jan 1st, 2012 and Jul 31st, 2025 will be retrospectively registered.
  Interventions: Other: Cardiac imaging

INTERVENTIONS:
Other: Cardiac imaging — Patients who underwent CTA or CAG, with or without other cardiac imaging modelities (OCT, IVUS, or CMR) will be enrolled in this registry.
  Other Names: CAG/CTA/OCT/IVUS/CMR

SUMMARY:
The purpose of this registry is to establish a multi-modality cardiac image database including coronary angiography (CAG), optical coherence tomography (OCT), intravascular ultrasound (IVUS), computed tomography angiograms (CTA) and cardiac magnetic resonance imaging (CMR) for future studies. The main goal of this collaboration is to create a resource for advanced research on atherosclerosis through image analysis.

DETAILED DESCRIPTION:
This registry plans to establish a multi-modality cardiac image database including coronary angiography (CAG), optical coherence tomography (OCT), intravascular ultrasound (IVUS), computed tomography angiograms (CTA) and cardiac magnetic resonance imaging (CMR) for future studies. Patients who underwent CAG or CTA during Aug 1st, 2025 and Dec 31st, 2035 at Zhongshan Hospital will be included in this registry. In addition, patients with CTA or at least one of OCT/IVUS/CMR between Jan 1st, 2012 and Jul 31st, 2025 will be retrospectively registered. Subgroups of these patients will have OCT/IVUS/CMR as according to their clinical presentations and requests from their doctors in charge. This registry aims to create a resource for advanced imaging research on atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with potential cardiovascular disease(s) (CVD) or diagnosed with CVD who were referred to CTA and/or CAG.
* Optional cardiac imagings, namely OCT/IVUS/CMR were up to doctors in charge and not mandatory.

Exclusion Criteria:

* Patient without any of the above mentioned cardiac imaging record.

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with potential cardiovascular disease(s) (CVD) or diagnosed with CVD who were referred to CTA and/or CAG at Zhongshan Hospital, Fudan university.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2045-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | 10 years
  Major adverse cardiac events

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, MD, PhD, Principal Investigator — Cardiovascular Department, Zhongshan Hospital, Fudan University

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD for this observational study.